CLINICAL TRIAL: NCT00075946
Title: Randomized Phase III Trial Comparing Two Different Rituximab Dosing Regimens For Patients With Low Tumor Burden Indolent Non-Hodgkin's Lymphoma
Brief Title: Rituximab in Treating Patients With Low Tumor Burden Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000346359; U10CA021115 (NIH); ECOG-E4402 (Other: Eastern Cooperative Oncology Group)
Record Dates: First submitted 2004-01-12; First posted 2004-01-14 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Rituximab Retreatment (Active Comparator): Patients receive rituximab IV once a week for 4 weeks upon disease progression provided time to progression is more than 6 months.
  Interventions: Biological: rituximab
- Arm B: Rituximab Scheduled (Experimental): Patients receive a single dose of rituximab IV once every 13 weeks until disease progression and in the absence of unacceptable toxicity.
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known which rituximab regimen is more effective in treating indolent non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two different schedules of rituximab and comparing them to see how well they work in treating patients with low tumor burden indolent stage III non-Hodgkin's lymphoma or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare time to rituximab failure between the rituximab scheduled and rituximab retreatment arms.

Secondary

* To compare the time to first cytotoxic therapy between the rituximab scheduled and rituximab retreatment arms.
* To document the rationale for beginning cytotoxic therapy; defined as chemotherapy, radiation therapy or radioimmunotherapy.
* To compare the toxicities associated with rituximab therapy between the two randomized treatment arms.
* Quality of Life Objectives:

  1. To compare health-related quality of life, distress, psychological functioning, physical well-being and functional well-being of patients receiving rituximab scheduled to those receiving rituximab retreatment.
  2. To examine the impact of differential treatment response (delayed time to rituximab failure and/or time to first cytotoxic therapy), if observed, on quality of life, distress, and psychological functioning on patients receiving rituximab scheduled to those receiving rituximab retreatment.
  3. To obtain prospective data on physical and functional well-being during treatment with rituximab.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to histologic subtype (follicular vs other), age (under 60 vs 60 and over), and the time from diagnosis (less than 1 year vs at least 1 year).

* Induction rituximab: Patients receive rituximab Intravenous (IV) once a week for 4 weeks.

Patients are re-evaluated 9 weeks after the completion of induction rituximab. Patients with a partial or complete response to induction rituximab are randomized to 1 of 2 treatment arms.

* Arm A (retreatment rituximab): Patients receive rituximab IV once a week for 4 weeks upon disease progression provided time to progression is more than 6 months.
* Arm B (scheduled rituximab): Patients receive a single dose of rituximab IV once every 13 weeks until disease progression and in the absence of unacceptable toxicity.

Quality of life is assessed after induction rituximab treatment and at 26, 39, 65, 117, 169, and 221 weeks after randomization.

Patients are followed at least annually for 15 years from study entry.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically confirmed non-Hodgkin's lymphoma, including 1 of the following:

  * Follicular grade 1 or 2
  * Small lymphocytic
  * Marginal zone (nodal)
  * Marginal zone (splenic)
  * Mucosa-associated lymphoid tissue (MALT)
* Stage III or IV disease
* Must meet the following criteria for low tumor burden:

  * No nodal or extranodal mass at least 7 cm
  * Less than 3 nodal masses greater than 3 cm in diameter
  * No systemic symptoms or B symptoms
  * No splenomegaly greater than 16 cm by a computed tomography (CT) scan
  * No evidence of risk of compression of a vital organ (i.e., ureteral or epidural)
  * No leukemic phase with greater than 5,000/mm^3 circulating lymphocytes
  * No cytopenias, defined as any of the following:

    * Platelet count less than 100,000/mm^3
    * Hemoglobin less than 10 g/dL
    * Absolute neutrophil count less than 1,500/mm^3
* At least 1 objective measurable disease parameter

  * Abnormal positron emission tomography (PET) scans will not constitute evaluable disease unless verified by CT scan or other appropriate imaging
* Age: 18 and over
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Must meet the following criteria for labs:

  * Hematopoietic

    * Absolute neutrophil count at least 1,500/mm^3*
    * Hemoglobin at least 10 g/dL*
    * Platelet count at least 100,000/mm^3*
    * NOTE: *Without growth factor and/or transfusion support
  * Hepatic

    * Bilirubin no greater than 2 times upper limit of normal (ULN) OR direct bilirubin normal for patients with Gilbert's Syndrome
    * The aspartate transaminase (AST) and alanine transaminase (ALT) ratio (AST/ALT) no greater than 5 times ULN
    * Hepatitis B surface antigen negative
  * Renal

    * Creatinine no greater than 2 times ULN

EXCLUSION CRITERIA:

* Evidence of transformation to a large cell histology
* Pregnant or nursing. Fertile patients must use effective contraception
* HIV positive
* Uncontrolled active infection
* Other malignancy within the past 2 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Prior immunotherapy for lymphoma
* Prior chemotherapy for lymphoma
* Concurrent chemotherapy
* Prior radiotherapy for lymphoma
* Concurrent radiotherapy
* Concurrent radioimmunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2004-01-23 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S. Kahl, MD, Study Chair — University of Wisconsin, Madison
Locations (483):
- United States (483):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Camino Medical Group - Treatment Center, Sunnyvale, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Johnson County Radiation Therapy, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - MaineGeneral Medical Center - Waterville, Waterville, Maine
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - Kaiser Permanente - Towson, Lutherville, Maryland
  - Kaiser Permanente Capital Area Medical Group - Shady Grove Facility, Rockville, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Morton Hospital & Medical Center, Taunton, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City Cancer Center at St. Joseph's Medical Mall, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Radiation Oncology Associates of Kansas City at Northland Radiation Oncology Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Carson Tahoe Cancer Center at Carson Tahoe Regional Medical Center, Carson City, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - AtlantiCare Cancer Care Institute at AtlantiCare Regional Medical Center - Mainland Campus, Pomona, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Underwood Memorial Hospital, Woodbury, New Jersey
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Richard G. Laube Cancer Center at ACMH, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Mountain Oncology Group, Bennington, Vermont
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Kaiser Permanente Medical Center - Fair Oaks, Fairfax, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Francis Hospital, Federal Way, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Kahl BS, Williams ME, Hong F, et al.: Preliminary pharmacokinetic (PK) analysis of Eastern Cooperative Oncology Group Protocol E4402: rituximab extended schedule or re-treatment trial (RESORT) . [Abstract] Blood 110 (11): A-3420, 2007.
- [Result] Kahl BS, Hong F, Williams ME, Gascoyne RD, Wagner LI, Krauss JC, Habermann TM, Swinnen LJ, Schuster SJ, Peterson CG, Sborov MD, Martin SE, Weiss M, Ehmann WC, Horning SJ. Rituximab extended schedule or re-treatment trial for low-tumor burden follicular lymphoma: eastern cooperative oncology group protocol e4402. J Clin Oncol. 2014 Oct 1;32(28):3096-102. doi: 10.1200/JCO.2014.56.5853. Epub 2014 Aug 25. PMID 25154829
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened on Nov 21, 2003, accrued its first patient on January 23, 2004, and closed on Sept 12, 2008, with final accrual of 545 patients.
Pre-assignment Details: Patients received induction rituximab IV once a week for 4 weeks. Patients were re-evaluated 9 weeks after the completion of induction rituximab. Patients with a partial or complete response to induction rituximab were randomized to one of the two treatment arms, stratified on histology (follicular vs other), age, and time from diagnosis.
Groups:
- Rituximab Retreatment: Follicular Patients; Rituximab Retreatment: Non-Follicular Patients: Following induction rituximab, patients who were randomized to this arm received rituximab IV once a week for 4 weeks upon disease progression provided time to progression is more than 6 months. Follicular and non-follicular patients were analyzed separately per protocol.
- Rituximab Scheduled: Follicular Patients; Rituximab Scheduled: Non-Follicular Patients: Following induction rituximab, patients who were randomized to this arm received a single dose of rituximab IV once every 13 weeks until disease progression and in the absence of unacceptable toxicity. Follicular and non-follicular patients were analyzed separately per protocol.
- Enrolled But Not Randomized: Patients who were enrolled in the study but not proceed to randomization. These could include patients with undetermined histology as well as those who did not achieve response (PR or CR) after induction rituximab.
Period: Overall Study
Arm/Group | Rituximab Retreatment: Follicular Patients | Rituximab Scheduled: Follicular Patients | Rituximab Retreatment: Non-Follicular Patients | Rituximab Scheduled: Non-Follicular Patients | Enrolled But Not Randomized
Started | 148 | 151 | 28 | 30 | 188
Treated and With Toxicity Data Available | 142 | 148 | 27 | 29 | 154
Included in Primary Analysis | 143 | 146 | 23 | 29 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 148 | 151 | 28 | 30 | 188
Not completed — Path ineligible: undetermined histology | 0 | 0 | 0 | 0 | 6
Not completed — Did not achieve response after induction | 0 | 0 | 0 | 0 | 182
Not completed — Incorrectly randomized (no response) | 5 | 5 | 5 | 1 | 0
Not completed — Adverse Event | 2 | 10 | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 58 | 4 | 9 | 0
Not completed — Alternative therapy | 16 | 2 | 5 | 0 | 0
Not completed — Other complicating disease | 7 | 13 | 1 | 4 | 0
Not completed — No response to retreatment | 23 | 0 | 2 | 0 | 0
Not completed — Time to progression less than 6 months | 15 | 30 | 8 | 3 | 0
Not completed — Other | 57 | 32 | 3 | 11 | 0

BASELINE CHARACTERISTICS:
Population: As the primary analysis only includes randomized patients, the baseline characteristics were provided among patients who were correctly randomized to one of the two arms for maintenance therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Retreatment: Follicular Patients | Rituximab Scheduled: Follicular Patients | Rituximab Retreatment: Non-Follicular Patients | Rituximab Scheduled: Non-Follicular Patients | Total
Number analyzed (Participants) | 143 | 146 | 23 | 29 | 341
Age, Continuous [Median (Full Range); unit: years] | 59 [25 to 86] | 58 [25 to 86] | 61 [47 to 86] | 65 [38 to 85] | 60 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 80 | 16 | 14 | 186
  Male | 67 | 66 | 7 | 15 | 155

OUTCOME MEASURES:

1. Primary Outcome: Time to Rituximab Failure (TTRF)
Description: TTRF is defined as the time from randomization until any one of the following criteria are met, and censored at last disease assessment for cases who have not experienced failure (with the cut-off date for final analysis of 11/1/2011): 1. No response (partial response (PR) or complete response (CR)) to rituximab retreatment (Arm A treatment). 2. Time to progression < 26 weeks from day 1 of most recent rituximab treatment. 3. Initiation of alternative therapy. 4. Inability to complete protocol therapy (due to adverse events, patient preference, or any other reason, including death).
Time Frame: Assessed (by restaging CT scans) 26 weeks ± 2 weeks from each rituximab treatment (including induction), counting the first rituximab dose as Day 1, until rituximab failure observed or July 17, 2013, whichever occurred first.
Population: Eligible patients who were randomized to one of the two arms for maintenance therapy.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Rituximab Retreatment: Follicular Patients | Rituximab Scheduled: Follicular Patients | Rituximab Retreatment: Non-Follicular Patients | Rituximab Scheduled: Non-Follicular Patients
Number analyzed (Participants) | 143 | 146 | 23 | 29
years | 3.92 [3.09 to 4.93] | 4.32 [3.53 to 4.98] | 1.39 [1.07 to NA] — Upper boundary has not been reached | 4.83 [2.46 to NA] — Upper boundary has not been reached
Statistical Analysis 1: Comparison: Rituximab Retreatment: Follicular Patients vs Rituximab Scheduled: Follicular Patients; The primary analysis is to compare the time to rituximab failure (TTRF) between the retreatment arm and the scheduled arm in follicular patients; Test type: Superiority or Other; p = 0.33, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.90 to 1.88] — Hazard ratio is for Rituximab Retreatment Arm/Rituximab Scheduled Arm in follicular patients
Statistical Analysis 2: Comparison: Rituximab Retreatment: Non-Follicular Patients vs Rituximab Scheduled: Non-Follicular Patients; Test type: Superiority or Other; p = 0.012, Log Rank; Hazard Ratio (HR) = 2.75, 95% CI 2-sided [1.22 to 6.19] — Hazard ratio is for Rituximab Retreatment Arm/Rituximab Scheduled Arm in non-follicular patients

2. Secondary Outcome: Time to First Cytotoxic Therapy (TTFC)
Description: TTFC is defined as the time from randomization to the time of first cytotoxic therapy (chemo and radio therapy), and censored as last follow-up time if no cytotoxic therapy has been used. Since median TTFC was not reached in 3 out of the 4 groups, 3-year TTFC was reported which was defined as the probability of not starting first cytotoxic therapy at 3 years.
Time Frame: Assessed every 13 weeks until rituximab failure observed or August 2013, whichever occurred first.
Population: Patients who were correctly randomized to one of the two maintenance arms.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Rituximab Retreatment: Follicular Patients | Rituximab Scheduled: Follicular Patients | Rituximab Retreatment: Non-Follicular Patients | Rituximab Scheduled: Non-Follicular Patients
Number analyzed (Participants) | 143 | 146 | 23 | 29
probability | 0.84 [0.78 to 0.90] | 0.95 [0.91 to 0.99] | 0.72 [0.55 to 0.94] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Rituximab Retreatment: Follicular Patients vs Rituximab Scheduled: Follicular Patients; Test type: Superiority or Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 3.21, 95% CI 2-sided [1.45 to 7.13] — Hazard ratio is for Rituximab Retreatment Arm/Rituximab Scheduled Arm in follicular patients
Statistical Analysis 2: Comparison: Rituximab Retreatment: Non-Follicular Patients vs Rituximab Scheduled: Non-Follicular Patients; Test type: Superiority or Other; p = 0.0002, Log Rank

3. Secondary Outcome: Overall Health-related Quality of Life (HRQL) at 6 Month After Randomization
Description: The overall HRQL was measured by the change in Functional Assessment of Cancer Therapy - General (FACT-G) from baseline to 6 months after randomization. The FACT-G is a 27-item assessment used to measure HRQL, specifically, physical, functional, social and emotional well-being. The total score ranges from 0 to 108, with higher scores indicating better HRQL.
Time Frame: Assessed at baseline and 6 months after randomization.
Population: Patients with patient-reported outcomes (PRO) data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm A: Rituximab Retreatment: Following induction rituximab, patients who were randomized to this arm received rituximab IV once a week for 4 weeks upon disease progression provided time to progression is more than 6 months.
- Arm B: Rituximab Scheduled: Following induction rituximab, patients who were randomized to this arm received a single dose of rituximab IV once every 13 weeks until disease progression and in the absence of unacceptable toxicity.
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Rituximab Scheduled
Number analyzed (Participants) | 128 | 125
units on a scale | 1.04 (12.82) | -0.71 (9.38)
Statistical Analysis 1: Comparison: Arm A: Rituximab Retreatment vs Arm B: Rituximab Scheduled; Test type: Superiority or Other; p = 0.270, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 10 years
Groups:
- Arm I: Induction Rituximab: Patients received rituximab IV once a week for 4 weeks. Patients were re-evaluated 9 weeks after the completion of induction rituximab. Patients with a partial or complete response to induction rituximab were randomized to one of the two treatment arms.
Arm/Group | Arm I: Induction Rituximab | Arm A: Rituximab Retreatment | Arm B: Rituximab Scheduled
Serious Adverse Events (participants affected / at risk) | 23/500 | 5/169 | 10/177
Other Adverse Events (participants affected / at risk) | 36/500 | 5/169 | 14/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Induction Rituximab (N=500) | Arm A: Rituximab Retreatment (N=169) | Arm B: Rituximab Scheduled (N=177)
Anaphylaxis (Immune system disorders) | 2 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 2 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 3
Fever (General disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Peripheral nerve infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, spe (Infections and infestations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 8 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Induction Rituximab (N=500) | Arm A: Rituximab Retreatment (N=169) | Arm B: Rituximab Scheduled (N=177)
Fatigue (General disorders) | 36 | 5 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No